CLINICAL TRIAL: NCT05812807
Title: OptimICE-PCR: De-Escalation of Therapy in Early-Stage TNBC Patients Who Achieve pCR After Neoadjuvant Chemotherapy With Checkpoint Inhibitor Therapy
Brief Title: Pembrolizumab vs. Observation in People With Triple-negative Breast Cancer Who Had a Pathologic Complete Response After Chemotherapy Plus Pembrolizumab
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A012103; NCI-2022-07859 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2023-03-23; First posted 2023-04-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Early Stage Triple-Negative Breast Carcinoma
MeSH Terms: interventions — pembrolizumab; Watchful Waiting; Observation; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV on study. Patients also undergo tumor biopsy on study, and collection of blood on study and during follow-up.
  Interventions: Biological: Pembrolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm II (observation) (Experimental): Patients undergo observation on study. Patients also undergo tumor biopsy on study, and collection of blood on study and during follow-up.
  Interventions: Other: Patient Observation; Procedure: Biopsy; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda
  Arms: Arm I (pembrolizumab)
Other: Patient Observation — Undergo observation
  Other Names: Active surveillance; watchful waiting; observation
  Arms: Arm II (observation)
Procedure: Biopsy — Undergo biopsy
Procedure: Biospecimen Collection — Undergo collection of blood
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
The phase III trial compares the effect of pembrolizumab to observation for the treatment of patients with early-stage triple-negative breast cancer who achieved a pathologic complete response after preoperative chemotherapy in combination with pembrolizumab. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. This trial may help researchers determine if observation will result in the same risk of cancer coming back as pembrolizumab after surgery in triple-negative breast cancer patients who achieve pathologic complete response after preoperative chemotherapy with pembrolizumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether observation results in a non-inferior recurrence-free survival (RFS) compared to adjuvant pembrolizumab in early-stage triple-negative breast cancer (TNBC) patients who achieve a pathologic complete response (pCR) after neoadjuvant chemotherapy with pembrolizumab.

II. To compare quality of life (QOL) at approximately 27 weeks as assessed by the Functional Assessment of Cancer Therapy-Breast (FACT-B) Trial Outcome Index between patients randomized to adjuvant pembrolizumab versus observation. (Quality of Life) III. To assess the social value of de-escalation of adjuvant breast cancer immunotherapy at approximately 27 weeks and, by modeling, over a lifetime. (Value of Care)

SECONDARY OBJECTIVES:

I. To evaluate whether observation compared to adjuvant pembrolizumab impacts the following:

Ia. RFS by stage at presentation and by receipt of prior anthracycline therapy; Ib. Adverse event rate: difference in Grade 3 or higher adverse event rates overall and Grade 3 or higher immune-related adverse events (irAEs) rates; Ic. Overall Survival (OS); Id. Locoregional recurrence (LRR both isolated LRR as first events and LRR events simultaneous with DM); Ie. RFS, LRR, OS, adverse events, and QOL by age (=< 45, 46-65, and > 65), race, and ethnicity; If. Adverse events related to receipt of radiotherapy. II. To assess the value of de-escalation of breast cancer immunotherapy from the payer perspective at approximately 27 weeks and, by modelling, over a lifetime. (Value of Care) III. To compare patient out-of-pocket costs at approximately 27 weeks between patients randomized to adjuvant pembrolizumab versus observation. (Value of Care) IV. To compare financial toxicity at approximately 27 weeks between patients randomized to adjuvant pembrolizumab versus observation. (Value of Care) V. To compare work/productivity impairment at approximately 27 weeks between patients randomized to adjuvant pembrolizumab versus observation. (Value of Care)

EXPLORATORY OBJECTIVES:

I. To describe trajectories of QOL over time among patients randomized to adjuvant pembrolizumab versus (vs.) observation. (Quality of Life) II. To compare various QOL domains after approximately 27 weeks as assessed by the 5 subscales of the FACT-B Index between patients randomized to adjuvant pembrolizumab versus observation. (Quality of Life) III. To compare self-reported symptomatic adverse events at approximately 27 weeks assessed by the patient reported outcome Common Terminology Criteria for Adverse Events (PRO-CTCAE) between patients randomized to adjuvant pembrolizumab versus observation. (Quality of Life) IV. To describe trajectories of financial toxicity and work/productivity impairment over time from baseline to approximately 27 weeks among patients randomized to adjuvant pembrolizumab versus observation. (Value of Care) V. To develop and assess a measure of value from the patient perspective at approximately 27 weeks. (Value of Care)

OUTLINE: Patients are randomized to 1 of 2 arms after completing neoadjuvant chemotherapy in combination with pembrolizumab, followed by definitive breast surgery.

ARM I (PEMBROLIZUMAB): Patients receive pembrolizumab intravenously (IV) on study. Patients also undergo tumor biopsy on study, and collection of blood on study and during follow-up.

ARM II (OBSERVATION): Patients undergo observation on study. Patients also undergo tumor biopsy on study, and collection of blood on study and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Triple Negative Breast Cancer:

  * Patients with a history of stage T1cN1-2 or T2-4N0-2 breast cancer according to the primary tumor-regional lymph node anatomic staging criteria of the American Joint Committee on Cancer (AJCC), 8th edition as determined by the investigator in radiologic assessment, clinical assessment or both
  * Patients must have no residual invasive disease in the breast or lymph nodes after the completion of neoadjuvant therapy. Residual ductal carcinoma in situ (DCIS) is allowed. Isolated tumor cells are considered node-negative
  * Estrogen (ER) and progesterone (PR) =< 10%; HER2-negative by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines (immunohistochemistry [IHC] and fluorescence in situ hybridization [FISH])
  * If invasive disease was present in both breasts, participation in the study is permitted as long as the eligibility criteria are met for both tumors/breasts
* Patients must have received neoadjuvant chemotherapy in combination with pembrolizumab for a minimum of 6 cycles. All systemic chemotherapy and ICI therapy should have been completed preoperatively
* An interval of no more than 12 weeks between the completion date of the final surgery and the date of randomization

  * Note: Adjuvant radiation can be given on study. If given, it is encouraged to be given concurrently with pembrolizumab, per investigator discretion. Treatment with adjuvant pembrolizumab is strongly discouraged prior to participation in this trial, but if administered (e.g., if patients are awaiting pathology results), pembrolizumab may be administered for up to 6 weeks post-surgery and must be completed prior to registration
* Use of investigational anti-cancer agents must be discontinued at time of registration
* Adequate excision: Surgical removal of all clinically evident disease in the breast and lymph nodes as follows:

  * Breast surgery: Total mastectomy or breast-conserving surgery with histologically negative margins, including no ink on tumor for DCIS, at the time of excision

    ** For patients who undergo breast-conserving surgery, the margins of the resected specimen must be histologically free of ductal carcinoma in-situ (DCIS) as determined by the local pathologist. If pathologic examination demonstrates DCIS at the line of resection, additional operative procedures may be performed to obtain clear margins. If DCIS is still present at the resected margin after re-excision(s), the patient must undergo total mastectomy to be eligible. Patients with margins positive for classic lobular carcinoma in situ (LCIS) are eligible without additional resection
  * Lymph node surgery:

    * For a patient with clinically N0 disease, a sentinel lymph node biopsy should have been performed at time of surgical evaluation, and if pathologically node positive, the patient is no longer eligible. Isolated tumor cells are considered node-negative
    * For a patient with clinically N1 disease at diagnosis (with positive results from a fine-needle aspiration, core biopsy, or sentinel node biopsy performed prior to preoperative therapy) additional surgical evaluation of the axilla following preoperative therapy is required

      *** If they become cN0 (no palpable adenopathy), then a sentinel lymph node biopsy could have been performed at time of surgery (axillary dissection would also be permitted); if the sentinel lymph node biopsy is positive, the patient is no longer eligible
    * If sentinel node biopsy performed before preoperative therapy was negative, no additional surgical evaluation of the axilla is required after preoperative therapy. If sentinel node biopsy performed before preoperative therapy was positive, an ALND is required after preoperative therapy
    * If the only sentinel node identified by isotope scan is in the internal mammary chain, surgical evaluation of the axilla is still required
    * If sentinel node evaluation after preoperative therapy is negative, no further additional surgical evaluation of the axilla is required
    * Axillary dissection without sentinel node evaluation is permitted as the initial or sole axillary evaluation after preoperative therapy
* If breast-conserving surgery was performed but patient will not be receiving breast radiation, the patient is not eligible
* Not pregnant and not nursing, because this study involves an agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative serum or urine pregnancy test done =< 7 days prior to randomization is required
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet Count >= 100,000/mm^3
* Estimated glomerular filtration rate (eGFR) >= 15 mL/min/1.73m^2
* Total Bilirubin =<1.5 x upper limit of normal (ULN)

  * Patients with Gilbert's disease with a total bilirubin =< 2.5 x ULN and direct bilirubin within normal limits are permitted
* Aspartate aminotransferase (AST) serum aspartate aminotransferase [SGOT] / alanine aminotransferase (ALT) serum glutamic pyruvic transaminase [SGPT] =< 3 x institutional ULN
* Patients must be willing to provide tumor tissue from the diagnostic core biopsy. If inadequate tumor tissue is available, patients are still eligible to participate in the trial
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial

Exclusion Criteria:

* No stage IV (metastatic) breast cancer
* No history of any prior (ipsi- or contralateral) invasive breast cancer. Prior DCIS is allowed
* No evidence of recurrent disease following preoperative therapy and surgery
* No known active liver disease, e.g. due to hepatitis B virus (HBV), hepatitis C virus (HCV), autoimmune hepatic disorders, or sclerosing cholangitis
* No history of intolerance, including Grade 3 or 4 infusion reaction or hypersensitivity to pembrolizumab or murine proteins or any components of the product

  * Note: Prior immune-related adverse events (irAEs) are allowed if they resolved and the patient tolerated subsequent therapy without requiring chronic steroids for the irAE
* No medical conditions that require chronic systemic steroids (>10 mg prednisone daily or equivalent) or any other form of immunosuppressive medications and has required such therapy in the last two years. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic therapy
* Patients who are unable or unwilling to comply with the requirements of the protocol per investigator assessment are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1295 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2033-05-31 (Estimated); Study Completion 2033-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | Up to 10 years.
  Defined as the time from randomization to first invasive local, regional, or distant recurrence or death due to any cause. RFS will be compared between treatment arms using the hazard ratio (with 90% confidence interval and stratified log-rank test) from a stratified Cox model.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 27 weeks after registration
  Adverse events will be determined using the latest version of the Common Terminology Criteria for Adverse Events (CTCAE). The proportions of patients with a grade 3 or higher AE will be compared between the arms using a chi-square test. A similar analysis will be done to compare the grade 3 or higher irAE rates
Overall survival | Up to 10 years.
  Defined as the time from randomization to death due to any cause. OS will be compared between treatment arms using the hazard ratio (and stratified log-rank test) from a stratified Cox model
Locoregional recurrence incidence | Up to 10 years.
  Defined as the time from randomization to first invasive local or regional recurrence. The cumulative incidence of LRR will be compared between treatment arms using a log-rank test (and estimated using Kaplan-Meier curves).
Radiation adverse events | Up to 27 weeks after registration
  Radiation adverse events include pneumonitis, hypothyroidism and dermatitis. Radiation AE event rates will be determined for patients who received radiation. The numerator is the number of patients with the radiation AE and the denominator is the number of patients who received radiation. The analysis of the radiation related adverse event rates will only include patients who received radiation treatment. The radiation AE rates will be compared between the two arms using a chi-square test.

CONTACTS AND LOCATIONS:
Locations (826):
- United States (809):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Marshall Cancer Center, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Enloe Medical Center, Chico, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Stanford Cancer Center Emeryville, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Mills Health Center, San Mateo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Schulze Family Foundation Cancer Clinic - Bonita Health Center, Bonita Springs, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Orlando Health Cancer Institute - Lake Mary, Lake Mary, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Health Central, Ocoee, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Mease Countryside Hospital, Safety Harbor, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MEJ, Council Bluffs, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Hamburg, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Tufts Medical Center Cancer Center Stoneham, Stoneham, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Mary Lanning Memorial Hospital, Hastings, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - The Philips Family Cancer Center, Southampton, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Cone Health Cancer Center at Asheboro, Asheboro, North Carolina
  - Cone Health MedCenter Asheboro, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Health Cancer Care Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - UNC Health Cancer Care Garner, Garner, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Levine Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Levine Cancer Institute - Union West, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Wakefield, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - OhioHealth O'Bleness Hospital, Athens, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Yolanda G Barco Oncology Institute, Meadville, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute - Mitchell, Mitchell, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Tarrant County Hospital District/JPS Health Network, Fort Worth, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Kaiser Permanente-Caton Hill Medical Center, Woodbridge, Virginia
  - FHCC Overlake, Bellevue, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Valley Medical Center, Renton, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (13):
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHU de Quebec-Hopital du Saint-Sacrement (HSS), Québec, Quebec
  - Centre Hospitalier Regional de Trois-Rivieres, Trois-Rivières, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Puerto Rico (4):
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Undecided